CLINICAL TRIAL: NCT03741582
Title: Urban Transformations and Health: the Case of TransMiCable in Bogotá
Acronym: TRUST
Status: Active, not recruiting | Type: Observational
Sponsor: University of Los Andes, Columbia (Other)
Collaborators: Wellcome Trust (Other); Drexel University (Other); Fundación Santa Fe de Bogota (Other)
Responsible Party: Principal Investigator, Olga Lucia Sarmiento, Professor, University of Los Andes, Columbia
Other Study IDs: 806-2017
Record Dates: First submitted 2018-10-19; First posted 2018-11-15 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Quality of Life; Social Capital; Transportation; Physical Activity; Homicide; Respiratory Disease
Keywords: Transportation; Urban Health; Quality of Life; Social Capital; Crime; Respiratory Diseases
MeSH Terms: conditions — Motor Activity; Respiration Disorders; Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control - San Cristobal: 1021 individuals located in an area with no access to the intervention (TransMicable). The control area was defined by a 800-meter buffer around each projected station of the car, "San Cristobal" was an area with a projected but non financed Cable Car.
- Intervention - Ciudad Bolviar: 1031 individuals who live in the area of influence of TransMiCable. The area of influence of TransMiCable was defined by a 800-meter radial buffer around each station of the cable car.
  Interventions: Other: TransMiCable

INTERVENTIONS:
Other: TransMiCable — TransMiCable will have one service line 3.43 km-long with four stations ("El Tunal" , "Juan Pablo II" , "Manitas" , and "Paraiso", see highlighted stops in Figure 2). "El Tunal" is the station that connects to the city's bus rapid transit system. The planned capacity of TransMiCable is 3,600 persons per hour in 163 cabins or gondolas. Each cabin fits ten passengers, with space for wheelchairs and bicycles and will be equipped with free Wi-Fi. The expected travel time reductions from each station to portal "El Tunal", through the shortest pathway, are: 26 minutes saved from "Juan Pablo II" station-from 32 to 6 minutes; 31 minutes saved from "Manitas" station-from 38 to 7 minutes and 49 minutes saved from "Paraiso" station-from 62 to 13 minutes 22. In conjunction with TransMiCable, urban projects will be implemented including the construction of parks, outdoor gyms, sport courts, community centers for children and older adults, a market, an administrative, and a tourism offices.
  Groups: Intervention - Ciudad Bolviar

SUMMARY:
Cable cars are means of transportation with urban mobility benefits for vulnerable populations living in areas with geographic barriers. Despite their popularity, there is no evidence of cable cars' potential health effects. TransMicable, located in "Ciudad Bolivar", Bogota, Colombia will open in late-2018 presenting an unprecedented opportunity to assess the health impacts and accessibility improvements. The investigators aim is to assess the effect of theTransMiCable implementation on social determinants of health (social capital, employment, crime, transport, microenvironment pollution, built environment), healthy behaviors (leisure and transport physical activity) and health outcomes (health-related quality of life, respiratory diseases and homicides).

The investigators are conducting a controlled quasi-experimental pre-post study with six elements: 1) The co-construction of a conceptual framework using a causal loop diagram with stakeholders of multiple sectors. 2) A (non-intervention - intervention) quantitative study of social capital, community participation, travel time, costs, demand, modal choice, physical activity and health-related quality of life using repeated in-person questionnaire, anthropometric measurements and physical activity using accelerometers. 3) A transport trajectory study in a subsample of the population of the quantitative study using a mobile application to track journeys. 4) A subsample of environment evaluations 5) Our Voice in the Neighborhood qualitative study to address the potential change in perceptions of the neighborhood using Citizen Science "by the people" involving the community and local public and private stakeholders and 6) A Secondary-data analysis of Crime and Respiratory diseases using time trends from official surveillance systems for homicides and acute respiratory diseases.

The investigators' main hypothesis are 1) There is an increase in the Social Capital and Quality of life indicators in the TransMicable target area after the implementation when compared to other neighborhoods without TransMiCable. 2) There is a significant decrease in travel time and cost for trips to downtown Bogota and an increase in the total number of trips for residents of "Ciudad Bolivar" neighborhoods with TransMiCable, after the implementation of TransMiCable when compared to other neighborhoods without TransMiCable in the locality of "San Cristobal". 3) There is a significant shift in modal choice for the resident of "Ciudad Bolivar" from informal transport service to the TransMiCable system with a positive association in terms of proximity to TransMiCable stations. 4) Most TransMiCable users are former informal bus transit and formal bus feeder users. While most users will access TransMiCable by walking, some living further from stations will take informal transport services to access to TransMiCable. 5) There is a reduction in the microenvironment pollution around the target area of TransMiCable when compared to the control area. 6) There is a change in the perception of the neighborhood for residents of the target area of TransMiCable when compared to the control area. 7) There is a significant decrease in the prevalence of homicides and acute respiratory diseases in the area of the TransMiCable implementation in comparison to the control area without TransMiCable. The results of this study will allow us to understand baseline dynamics, while, in the long-term, allowing us to assess the changes in travel and health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Has minimum 18 years old
* Has lived over the past 2 years in the study area
* Would not move from the study area in the next 2 years
* Has not any kind of cognitive problem

Exclusion Criteria:

* Has less than 18 years old
* Has not lived over the past 2 years in the study area
* Has plans to move from the study area in the next 2 years
* Has any kind of cognitive problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Every participant of the study is an adult that lives on one of the 225 blocks selected from each buffer with probability proportional to the size of the catchment areas' population. For selecting the participant, 4 or 5 households were systematically selected on each block. The families of each household were selected with a random numbers chart, as well as the participant listing every adult by age.
Sampling Method: Probability Sample
Enrollment: 2052 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Basic activity monitoring | First measurement: February to December 2018, Second measurement: July 2019 to March 2020, Third measurement: March to Sep 2021, Fourth measurement: August 2022 to May 2023
  An Actigraph activity monitor is given to every participant of the study for wearing it over seven days. The reception of the monitors by the participants was prioritized in the intervention group over the control, due to the limited amount of monitors. Participants are asked to wear an ActiGraph "GT3X" or "GT3X+" accelerometer at the waist, and positioned in line with the right mid-axillary line, for at least seven consecutive days (plus an initial familiarization day and the morning of the final day) during all waking hours. Accelerometers are initialized to collect data at 60-second epochs. Participants who successfully complete the use of the monitor are included on a raffle for an special prize at the end of every measurement. In every follow-up participants will be asked to repeat the activity monitoring along with the questionnaire.
Trajectory measurement | First measurement: February to December 2018, Second measurement: July 2019 to March 2020, Third measurement: March to Sep 2021, Fourth measurement: August 2022 to May 2023
  We recorded the trajectories of a subset of participants using a global positioning system (GPS) mobile application. For the first measurement, the mobile phone application Moves was installed in participants' Smart-phones to automatically record an activity diary. The application remains installed for at least seven consecutive days (plus an initial familiarization day and the morning of the final day). Data produced by the mobile application include geo-location of places visited, departures and arrival times for each place, transportation modes used classified as walking, cycling, running, and motorized transport, and depending on the Smart-phone, routes employed to access to each destination with geo-located checkpoints. Since Moves servers shut down on july 31, for the follow-up measurements will use another GPS trajectory mobile application.
Longitudinal qualitative interviews | First measurement: February to December 2018, Second measurement: July 2019 to March 2020, Third measurement: March to Sep 2021, Fourth measurement: August 2022 to May 2023
  Our Voice in the Neighborhood qualitative study to address the potential change in perceptions of the neighborhood using Citizen Science "by the people" involving the community and local public and private stakeholders.
Questionnaire survey Transport section | First measurement: February to December 2018, Second measurement: July 2019 to March 2020, Third measurement: March to Sep 2021, Fourth measurement: August 2022 to May 2023
  Characterization of the use of public transport measured with questions taken from the Mobility Survey of Bogotá.
Questionnaire survey IPAQ section | First measurement: February to December 2018, Second measurement: July 2019 to March 2020, Third measurement: March to Sep 2021, Fourth measurement: August 2022 to May 2023
  Leisure-time physical activity spent time during a week measured with the International Physical Activity Questionnaire (IPAQ) in its long version.
Questionnaire survey Quality of life section | First measurement: February to December 2018, Second measurement: July 2019 to March 2020, Third measurement: March to Sep 2021, Fourth measurement: August 2022 to May 2023
  Quality of life and wellbeing measured with the World Health Organization Quality Of Life instrument (WHOQOL-bref instrument). The instrument produces a quality of life profile with a 26-item questionnaire divided in four domains: domains: physical health, psychological, social relationships and environment. It is possible to derive a score for each one of them, which denotes the individual perception of the quality of life in each component. The score goes from 0 and increases positively until 5 for each question being 5 the best outcome possible. The mean score of each domain is used for calculating the average score, and then multiplied by 4 for making the scores comparable with WHOQOL-100 (long version of the questionnaire).
Questionnaire survey Social capital section | First measurement: February to December 2018, Second measurement: July 2019 to March 2020, Third measurement: March to Sep 2021, Fourth measurement: August 2022 to May 2023
  Social Capital measured by an adapted questionnaire based on: The World Bank (SC-IQ), The Development Bank of Latin America - CAF survey, and Encuesta Multipropósito.
Questionnaire survey Respiratory diseases section | First measurement: February to December 2018, Second measurement: July 2019 to March 2020, Third measurement: March to Sep 2021, Fourth measurement: August 2022 to May 2023
  Identification of acute and chronic respiratory diseases in all the infants and elders in a household measured with a module of "less than 5" and "more than 65 years old"
Questionnaire survey loneliness section | First measurement: February to December 2018, Second measurement: July 2019 to March 2020, Third measurement: March to Sep 2021, Fourth measurement: August 2022 to May 2023
  Loneliness of the participant measured with the University of California, los Angeles (UCLA) Scale of Loneliness.
Questionnaire survey Use of free time section | First measurement: February to December 2018, Second measurement: July 2019 to March 2020, Third measurement: March to Sep 2021, Fourth measurement: August 2022 to May 2023
  An inventory of activities during free time, the time participants spend going to health, educational and recreational services, and whether during the last 12 months participants attended to preventive health services.
Environment evaluations SOPARC | First measurement: February to December 2018, Second measurement: July 2019 to March 2020, Third measurement: March to Sep 2021, Fourth measurement: August 2022 to May 2023
  Observed levels of physical activity in the parks and recreation centers using System for Observing Play and Recreation in Communities (SOPARC).
Environment evaluations Air pollution | First measurement: February to December 2018, Second measurement: July 2019 to March 2020, Third measurement: March to Sep 2021, Fourth measurement: August 2022 to May 2023
  personal exposure in transport microenvironments to fine particulate matter (PM2.5), equivalent black carbon (eBC), Carbon Monoxide (CO) and number of sub-micron particles (Np) using aerosol monitors, aethalometers and photoradiometers while keeping records of their time and activity while in the microenvironments.
Crime measurements | This measurements are performed by different official systems and were collected by the end of each year.
  A Secondary-data analysis of Crime using time trends from official surveillance systems for homicides.
Respiratory diseases measurements | This measurements are performed by different official systems and were collected by the end of each year.
  A Secondary-data analysis of Respiratory diseases using time trends from official surveillance systems for acute respiratory diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Olga L Sarmiento, Principal Investigator — Universidad de los Andes, Colombia
Locations (1):
- Universidad de los Andes, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: Undecided